CLINICAL TRIAL: NCT00141258
Title: Pregabalin Add-On Titration Trial: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of Pregabalin (150 mg - 600 mg/Day) Using a Flexible, Optimized Dose Schedule in Subjects With Partial Seizures
Brief Title: Pregabalin Epilepsy Add-On Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081079
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2009-04

CONDITIONS: Partial Seizures
MeSH Terms: conditions — Seizures | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin

SUMMARY:
To evaluate the efficacy of pregabalin as adjunctive therapy, using a flexible, optimized dose schedule with dose adjustment based on clinical response and tolerability, compared to placebo in subjects with partial seizures

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of epilepsy with partial seizures (as defined in the ILAE Classification of Seizures) and be currently taking 1-3 AEDs
* Have a minimum of 4 partial seizures occurring over at least 2 days during the 6-week baseline with no 28-day period free of partial seizures

Exclusion Criteria:

* Have a treatable cause of seizures
* Are currently receiving treatment with CNS-active compounds (exception: single antidepressant, hypnotics, and standard AEDs), vigabatrin, Felbatol (felbamate), Neurontin (gabapentin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2005-10; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Response ratio (RRatio or symmetrized percent change) for all partial seizures

SECONDARY OUTCOMES:
Responder rate, Percent change, Percent of SGTC responders, Seizure freedom measures, Change in number of seizure-free days (SFD) per a 28-day period, Analysis by seizure type, HADS, Weekly and endpoint mean sleep interference scores from DSIS, QOLIE-31

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- South Korea (5):
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081079&StudyName=Pregabalin+Epilepsy+Add%2DOn+Trial